CLINICAL TRIAL: NCT06392113
Title: Developing a Falls Management Tool for Adults With Intellectual Disabilities- Proof of Concept Study
Brief Title: Developing a Falls Management Tool for Adults With ID-POC
Status: Recruiting | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 22AS002
Record Dates: First submitted 2024-04-22; First posted 2024-04-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Intellectual Disability; Fall
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adults with an intellectual disability: Completion of ACTION FALLS programme
  Interventions: Behavioral: ACTION FALLS
- Carers of adults with an intellectual disability: Completion of ACTION FALLS programme
  Interventions: Behavioral: ACTION FALLS
- Clinicians working with adults with an intellectual disability: Completion of ACTION FALLS programme
  Interventions: Behavioral: ACTION FALLS

INTERVENTIONS:
Behavioral: ACTION FALLS — Falls prevention advice including booklet and videos

SUMMARY:
Falls can have a significant impact on the lives of adults with intellectual disabilities. The ACTION FALLS programme is a systematic falls management intervention that has been shown to be of benefit for older people however this programme in its current form needs to be adapted for use with adults with intellectual disabilities who have specific risk factors for falling and specific actions to reduce these risks. An adapted version of the programme to account for the different needs of adults with intellectual disabilities and the different services and support networks they access will be developed. A draft programme has been developed based on the views of adults with learning disabilities, carers and clinicians. This programme will now be tried out to see how easy it is to use and whether it can identify the falls risk factors relevant to adults with learning disabilities. Adults with an intellectual disability, clinicians and carers will t try out the programme and will be observed using it and will be asked to give verbal feedback on their views on how easy it is to complete and what could be improved.

DETAILED DESCRIPTION:
The draft ACTION FALLS programme that will be used in this proof-of-concept study includes the following sections:

* Section One: A falls checklist, videos, and resource booklet for adults with an ID and carers.
* Section Two: A falls checklist for clinicians and a clinician manual for use in a clinical service.

Section one has been designed to be able to be used by adults with an ID and their carers independently of a clinical service. Additionally, section one could be used to support a clinical assessment in a clinical team to capture the views of adults with an ID. Section two has been designed to be used by a healthcare professional undertaking a more detailed assessment with adults with an ID.

There will be two components of work to explore views and acceptability of both the sections of the programme and how they work independently and together.

Component One:

Up to 10 clinicians will be recruited, to collect data with up to 15 adults with ID. The clinicians will be working in the ID service within Nottinghamshire Healthcare NHS Foundation Trust and will be asked to use the updated ACTION FALLS programme with adults with an ID accessing this service who give consent. The 'Think Aloud' method will be used to explore the views of the adult with ID and clinician in using the programme. The programme will be completed in addition to the standard clinical assessment and at a separate time convenient to both the clinician and participant. Completion of this programme will not interfere with the standard care received by the participant and clinical care will remain the responsibility of the usual care team and existing processes.

The following data will be collected and analysed:

* Researcher field notes observing the completion of the programme. This will include the time taken to complete the programme and any barriers and facilitators (analysed thematically)
* Research field notes on the verbal feedback given by participants when completing the programme (analysed thematically)
* Completed programme (personal information will be removed by the researcher) - the number and type of risk factors identified will be extracted (analysed using descriptive statistics and themes)

Component Two:

Up to 15 adults with an ID and 5 carers supporting adults with an ID in Nottinghamshire will be asked to use section one of the programme. This will be done without any clinician involvement. The programme will be completed as part of the workshop.

The following data will be collected and analysed:

* Researcher field notes observing the participants using the programme, this will include the time taken to complete the checklist and any barriers and facilitators (analysed thematically). These will be anonymous.- Research field notes on the verbal feedback given by participants when reviewing the programme (analysed thematically). These will be anonymous.
* Completed programme (personal information will be removed by the clinical researcher) - the number and type of risk factors identified will be extracted (and analysed using descriptive statistics and themes).

Email addresses of participants who would like to be provided with a lay summary at the end of the study will be collected. This will be collected on the consent form optionally.

ELIGIBILITY:
Inclusion Criteria:

Component One:

* Adults with ID, 18 years and over, accessing the ID service in identified clinical team
* Clinicians working in identified clinical team for adults with ID

Component Two:

Adults with an ID, 18 years and over, living in Nottinghamshire Family or paid carer of an adult with an ID living in Nottinghamshire

Exclusion Criteria:

* Lack of capacity to provide informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with ID and clinicians working in an identified ID service in one locality in the UK and adults with ID and their carers identified from one geographical location in the UK.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-28 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
The number and types of falls risks identified | Through study completion, on average one month
  The number and types of falls risks identified
Time taken and level of completion of the programme | Through study completion, on average one month
  Time taken and level of completion of the programme
Barriers and facilitators to completing the programme | Through study completion, on average one month
  Barriers and facilitators to completing the programme

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Nottinghamshire Healthcare NHS Foundation Trust, Nottingham

IPD SHARING:
Plan to Share IPD: No
No individual sharing of participant data.

REFERENCES:
- See also: Study website — https://www.nottingham.ac.uk/research/groups/communityrehabilitation/projects/falls-management-programme/developing-a-falls-management-programme-for-adults-with-intellectual-disabilities.aspx